CLINICAL TRIAL: NCT01159912
Title: A Randomised, Double-blind, Double-dummy, Placebo Controlled (With Rescue Medication), Multicenter Study to Evaluate the Efficacy and Safety of Fluticasone Furoate Inhalation Powder in the Treatment of Persistent Asthma in Adults and Adolescents.
Brief Title: Evaluating the Efficacy and Safety of Fluticasone Furoate Inhalation Powder in the Treatment of Asthma in Adults and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112059
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Asthma
Keywords: fluticasone propionate; Fluticasone furoate
MeSH Terms: conditions — Asthma | interventions — Fluticasone; fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluticasone Furoate OD and Placebo BID (Experimental): Fluticasone furoate inhalation powder once daily and placebo inhalation powder twice daily for 24 weeks
  Interventions: Drug: Fluticasone furoate; Drug: Placebo
- Fluticasone Propionate BID and Placebo OD (Active Comparator): Fluticasone propionate inhalation powder twice daily and placebo inhalation powder once daily for 24 weeks
  Interventions: Drug: Fluticasone propionate; Drug: Placebo
- Placebo only BID (Placebo Comparator): Placebo inhalation powder twice daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate — Fluticasone propionate inhalation powder, 250 µg
  Arms: Fluticasone Propionate BID and Placebo OD
Drug: Fluticasone furoate — Fluticasone furoate inhalation powder, 100 µg
  Arms: Fluticasone Furoate OD and Placebo BID
Drug: Placebo — Placebo inhalation powder

SUMMARY:
A randomised, double-blind, double-dummy, placebo controlled (with rescue medication), multicenter study to evaluate the efficacy and safety of Fluticasone Furoate inhalation powder in the treatment of persistent asthma in adults and adolescents.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, double-dummy, parallel-group study to compare the efficacy and safety of Fluticasone Furoate Inhalation Powder 100mcg once daily and Fluticasone Propionate Inhalation Powder 250mcg twice daily with Placebo. Subjects will participate in the study for up to a maximum of 29 weeks (including screening, treatment and follow-up contact). The primary endpoint consists of change from baseline in clinic visit trough (pre-bronchodilator and pre-dose) FEV1 at the end of the 24 week treatment period. The nominated powered secondary endpoint is the change from baseline in the percentage of rescue-free 24 hour periods during the 24-week treatment period. Safety assessments include adverse events, oropharyngeal examinations, clinical chemistry and urine cortisol excretion. For subjects who have consented for pharmacogenetics, a blood sample will also be taken for pharmacogenetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Outpatient at least 12 years of age
* Both genders; females of child bearing potential must be willing to use approved birth control method
* Pre-bronchodilator FEV1 of 40-90% predicted
* Reversibility FEV1 of at least 12% and 200mLs
* Current asthma therapy that includes an inhaled corticosteroid for at least 4 weeks prior to first visit

Exclusion Criteria:

* History of life threatening asthma
* Respiratory infection or candidiasis
* Asthma exacerbation within 6 months prior to first visit
* Concurrent respiratory disease or other disease that would confound study participation or affect subject safety
* Allergies to study drugs, study drug excipients, medications related to study drugs
* Taking another investigational medication or medication prohibited for use during this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2010-06-30; Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (69):
- United States (48):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Green Valley, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Cutler Bay, Florida
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Shiloh, Illinois
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Franklin, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Collegeville, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Richmond, Virginia
- Belgium (4):
  - GSK Investigational Site, Gozée
  - GSK Investigational Site, Halen
  - GSK Investigational Site, Natoye
  - GSK Investigational Site, Tremelo
- Germany (9):
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Schwedt, Brandenburg
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Erfurt, Thuringia
  - GSK Investigational Site, Schmölln, Thuringia
  - GSK Investigational Site, Berlin
- Poland (6):
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Łomża
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 112059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant received treatment (placebo) but was not randomized. Thus, 350 participants were enrolled in the study; however, only 349 were randomized.
Pre-assignment Details: Participants (par.) meeting all inclusion criteria/no exclusion criteria during Visit 1 entered a 4-week Run-in Period (RIP). At Visit 2 (end of RIP), par. meeting the eligibility criteria were randomized to the 24-week Double blind Treatment Period. 1036 par. were screened, 349 were randomized, and 343 received >=1 dose of study treatment.
Groups:
- Placebo: Participants received placebo via a dry powder inhaler (DPI) once daily (OD) in the evening and placebo via the DISKUS/ACCUHALER twice daily (BID) for 24 weeks (168 days). In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- FF 100 µg OD: Participants received fluticasone furoate (FF) 100 microgram (µg) inhalation powder via a DPI OD in the evening plus placebo via the DISKUS/ACCUHALER BID for 24 weeks (168 days). In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- FP 250 µg BID: Participants received fluticasone propionate (FP) 250 µg BID via the DISKUS/ACCUHALER plus placebo via a DPI OD in the evening (total daily dose of 500 µg) for 24 weeks (168 days). In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
Period: Overall Study
Arm/Group | Placebo | FF 100 µg OD | FP 250 µg BID
Started | 115 | 114 | 114
Completed | 75 | 92 | 88
Not Completed | 40 | 22 | 26
Not completed — Adverse Event | 2 | 2 | 3
Not completed — Lack of Efficacy | 23 | 15 | 14
Not completed — Protocol Violation | 1 | 2 | 3
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Withdrawal by Subject | 10 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FF 100 µg OD | FP 250 µg BID | Total
Number analyzed (Participants) | 115 | 114 | 114 | 343
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (17.68) | 40.1 (16.17) | 41.4 (15.64) | 40.6 (16.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 63 | 72 | 203
  Male | 47 | 51 | 42 | 140
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage (HER) | 23 | 22 | 19 | 64
  Central/South Asian Heritage | 1 | 0 | 1 | 2
  Japanese/East Asian HER/South East Asian HER | 1 | 1 | 1 | 3
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 1
  White | 88 | 90 | 92 | 270
  American Indian or Alaska Native & White | 1 | 0 | 0 | 1
  Missing | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Clinic Visit Trough Evening (Pre-bronchodilator and Pre-dose) Forced Expiratory Volume in One Second (FEV1) at the End of the 24 Week Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is defined as the clinic visit (pre-bronchodilator and pre-dose) FEV1 measurement taken at the clinic visit at the end of the dosing interval. Pre-dose and pre-rescue albuterol/salbutamol trough FEV1 was measured electronically by spirometry in the evening at the Baseline through Week 24 clinic visits. The highest of 3 technically acceptable measurements was recorded. Baseline was the pre-dose value obtained at Visit 2. Change from Baseline was calculated as the Week 24 value minus the Baseline value. Analysis was performed using analysis of covariance (ANCOVA) with covariates of Baseline, region, sex, age, and treatment. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement at scheduled clinic visits was used to impute the missing measurements.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study medication. Only those participants with non-missing covariates and a post-Baseline FEV1 measurement were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 100 µg OD | FP 250 µg BID
Number analyzed (Participants) | 113 | 111 | 107
Liters | 0.015 (0.0394) | 0.161 (0.0398) | 0.159 (0.0406)
Statistical Analysis 1: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.009, ANCOVA; Mean Difference (Final Values) = 0.146, 95% CI 2-sided [0.036 to 0.257]
Statistical Analysis 2: Comparison: Placebo vs FP 250 µg BID; Test type: Superiority or Other; p = 0.011, ANCOVA; Median Difference (Final Values) = 0.145, 95% CI 2-sided [0.033 to 0.257]

2. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour (hr) Periods at the End of the 24-week Treatment Period
Description: The number of inhalations of rescue bronchodilator, albuterol/salbutamol inhalation aerosol, used during the day and night was recorded by the participants in a daily electronic diary (eDiary). Similarly, asthma symptoms were recorded in a daily eDairy by the participants every day in the morning and evening before taking any rescue or study medication and before the peak expiratory flow measurement. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered to be rescue free. The Baseline value was derived from the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | Placebo | FF 100 µg OD | FP 250 µg BID
Number analyzed (Participants) | 114 | 112 | 113
Percentage of rescue-free 24-hr periods | 6.5 (2.82) | 21.3 (2.85) | 24.3 (2.83)

3. Secondary Outcome: Mean Change From Baseline in Daily Trough Evening (PM) Peak Expiratory Flow (PEF) Averaged Over the First 12 Weeks and 24 Weeks of the 24-week Treatment Period
Description: PEF is a measure of lung function and is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning and evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Trough evening PEF is the PM PEF measured approximately 24 hours after the last evening administration of study drug. Change from Baseline (defined as the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily trough PM PEF over 12 weeks and 24 weeks of the 24-week Treatment Period (at Weeks 12 and 24) minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | Placebo | FF 100 µg OD | FP 250 µg BID
Number analyzed (Participants) | 114 | 112 | 112
Liters/minute (L/min)
  PM PEF, Week 1 to 12 | 0.4 (3.25) | 2.2 (3.28) | 4.8 (3.28)
  PM PEF, Week 1 to 24 | -1.3 (3.36) | 1.5 (3.39) | 4.3 (3.40)

4. Secondary Outcome: Mean Change From Baseline in Daily Morning (AM) PEF Averaged Over the First 12 Weeks and 24 Weeks of the 24-week Treatment Period
Description: PEF is a measure of lung function and is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning and evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline (defined as the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily AM PEF over 12 weeks and 24 weeks of the 24-week Treatment Period (at Weeks 12 and 24) minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | Placebo | FF 100 µg OD | FP 250 µg BID
Number analyzed (Participants) | 114 | 112 | 113
Liters/minute (L/min)
  AM PEF, Week 1 to 12 | 5.7 (3.41) | 13.2 (3.44) | 9.4 (3.43)
  AM PEF, Week 1 to 24 | 5.0 (3.45) | 13.9 (3.48) | 9.9 (3.47)

5. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour (hr) Periods at the End of the 24-week Treatment Period
Description: The number of inhalations of rescue bronchodilator, albuterol/salbutamol inhalation aerosol, used during the day and night was recorded by the participants in a daily electronic diary (eDiary). Similarly, asthma symptoms were recorded in a daily eDairy by the participants every day in the morning and evening before taking any rescue or study medication and before the peak expiratory flow measurement. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered to be symptom free. The Baseline value was derived from the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | Placebo | FF 100 µg OD | FP 250 µg BID
Number analyzed (Participants) | 114 | 112 | 113
Percentage of symptom-free 24-hr periods | 10.4 (2.77) | 19.3 (2.79) | 19.2 (2.78)

6. Secondary Outcome: Change From Baseline in the Total Asthma Quality of Life Questionnaire (AQLQ) (+12) Score at Week 12 and Week 24
Description: The AQLQ is a disease-specific, self-administered quality of life questionnaire used to evaluate the impact of asthma treatments on the quality of life of asthma sufferers. The AQLQ for 12 years and older (AQLQ [+12]) is a modified version of the AQLQ for use in asthma patients between the ages of 12 and 70. The AQLQ contains 32 items in 4 domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items), and environmental stimuli (4 items). For the 32 items on the questionnaire, the response format consists of a seven-point scale, where a value of 1 indicates "total impairment" and a value of 7 indicates "no impairment." The AQLQ total score is defined as the average of the scores from all 32 questions; thus, the total score ranges from 1 (indicates "total impairment") to 7 (indicates "no impairment"). Baseline was the total score obtained at Visit 3. Change from Baseline was calculated as the total score at Weeks 12 and 24 minus the total score at Baseline.
Time Frame: Baseline, Week 12, and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FF 100 µg OD | FP 250 µg BID
Number analyzed (Participants) | 115 | 114 | 114
Scores on a scale
  Week 12, n=85, 99, 99 | 0.45 (0.078) | 0.69 (0.072) | 0.73 (0.073)
  Week 24, n=74, 90, 86 | 0.51 (0.090) | 0.84 (0.082) | 0.67 (0.084)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the treatment period (up to Week 24).
Description: An on-therapy AE or SAE is defined as an AE with an onset on or after the start date of study medication, but not later than one day after the last date of study medication. SAEs and AEs were collected in members of the ITT Population, comprised of all participants randomized to treatment, who received at least one dose of study medication.
Arm/Group | Placebo | FF 100 µg OD | FP 250 µg BID
Serious Adverse Events (participants affected / at risk) | 2/115 | 4/114 | 1/114
Other Adverse Events (participants affected / at risk) | 30/115 | 37/114 | 19/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | FF 100 µg OD (N=114) | FP 250 µg BID (N=114)
Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Abscess (Infections and infestations) | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Epididymal cyst (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | FF 100 µg OD (N=114) | FP 250 µg BID (N=114)
Bronchitis (Infections and infestations) | 7 | 8 | 4
Nasopharyngitis (Infections and infestations) | 6 | 9 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 7 | 6
Pharyngitis (Infections and infestations) | 4 | 5 | 2
Sinusitis (Infections and infestations) | 1 | 4 | 2
Urinary tract infection (Infections and infestations) | 4 | 1 | 0
Headache (Nervous system disorders) | 5 | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.